CLINICAL TRIAL: NCT06225479
Title: PRescription Exercise for Older Men With Urinary Disease (PROUD) Pilot Study
Brief Title: PRescription Exercise for Older Men With Urinary Disease
Acronym: PROUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); University of California, San Diego (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DK135804-01 (NIH); R01DK135804 (NIH)
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: physical fitness; endurance training; resistance training; prostatism; male urogenital diseases; urinary bladder outlet obstruction; skeletal muscle; mitochondria
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Prostatism; Male Urogenital Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-center 2-arm pilot randomized control trial (RCT) of a 12-week remote exercise intervention and a health education control among 68 physically inactive older men with LUTS/BPH.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This will be a 2-arm, partially-blinded, attention-controlled RCT. The randomization scheme will be computer-generated by the study statistician without participant contact. Participants will be randomized 1:1 in randomly permuted block sizes (2 or 4) to the exercise intervention or health education control arm stratified by recruitment site and any BPH medication use (yes/no). The randomization scheme is uploaded to University of California San Francisco (UCSF) REDCap and the study coordinator will randomize participants in UCSF REDCap. Assessors (for urinary and physical function testing), data analysts, and investigators will remain blinded to participants' randomization arm.
  Primary outcomes will be collected using self-administered questionnaires without risk of unblinding. Intervention status and any variables related to intervention status will be recorded and stored in a separate database by unblinded Clinical Research Coordinator (CRC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Participants in this study arm will receive a remote health education program which consists of twice-monthly "Successful Aging" newsletters and phone calls to reinforce and discuss topics in each newsletter.
  Interventions: Other: Calls and Newsletter
- Exercise Arm (Experimental): Participants in this study arm will receive an individualized 12-week exercise intervention plus a remote health education program.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — An individualized 12-week exercise intervention that will follow American College of Sports Medicine guidelines to ensure a gradual safe increase in frequency and intensity. The exercise goals for participants in the intervention arm are to increase minutes/week of aerobic exercise, build strength and muscle mass, and improve flexibility, core strength, and balance progressively over the course of 12 weeks. The participants are prescribed 3 sessions of aerobic exercise lasting 45-75 minutes each, including warm up and cool down; 2 resistance training sessions per week, and at least 3 flexibility and balance sessions per week.
  Intervention arm receives the following: Control arm "Successful Aging" newsletter plus additional educational materials related to exercise, heart rate monitor and resistance bands, and two 90-minute sessions and ten 30-minute phone sessions over 12 weeks with an exercise coach (the first two sessions include a resistance training session).
  Arms: Exercise Arm
Other: Calls and Newsletter — A 12-week remote health education program developed by the study team to provide a control for the exercise intervention. Participants in this arm will receive a summary of the American College of Sports Medicine guidelines (self-directed and time-based), a twice-monthly "Successful Aging" newsletter with suggestions for health diet, stress reduction, and social engagement, and twice-monthly phone calls to reinforce and discuss topics in the newsletter and to review adverse events and change in medications.
  Arms: Control Arm

SUMMARY:
This is a single-center pilot randomized controlled trial among 68 physically "inactive" older men with lower urinary tract symptoms (LUTS) attributed to benign prostatic hyperplasia (LUTS/BPH) assessing a 12-week remote exercise intervention versus health education control.

DETAILED DESCRIPTION:
This study will provide valuable insights into the feasibility of an individualized, remotely-monitored, and home-based exercise intervention as well as the effect of this intervention on lower urinary tract symptom (LUTS) severity and mechanistic measures (physical function, lower urinary tract function, frailty-related mechanistic biomarkers) in a diverse group of older men with LUTS attributed to benign prostatic hyperplasia (BPH). The potential public health benefit to society in this study could be large, as the investigators are targeting a common condition in older men (one in three older men develop LUTS in their lifetime).

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or older.
2. Male sex at birth.
3. Moderate-to-severe LUTS over the past month (defined as International Prostate Symptom Score [IPSS] >=12).
4. A clinical diagnosis of LUTS/BPH as demonstrated by a current or prior BPH medication prescription (alpha-blocker, 5alpha-reductase inhibitor, daily phosphodiesterase type 5 inhibitor) OR untreated LUTS/BPH and a maximum urinary flow rate <=12 ml/sec.
5. Physically inactive as defined in the Molecular Transducers of Physical Activity Consortium (MoTrPAC): no more than 1 day per week, lasting no more than 60 minutes, of regular endurance/aerobic exercise [e.g., brisk walking, jogging, running, cycling, elliptical, or swimming activity that results in feelings of increased heart rate (HR), rapid breathing, and/or sweating] or resistance exercise [resulting in muscular fatigue] in the past year). Leisure walkers are eligible unless they meet the HR, breathing, and sweating criteria.
6. Able to walk 400m without sitting, leaning, or the help of another person (observed during exercise testing) to ensure safety while exercising with remote monitoring. Use of a straight cane is allowed.
7. Able to speak and complete questionnaires in English.
8. Have an iOS or Android smartphone capable of installing the Polar Beat app.

Exclusion Criteria:

1. Prescribed overactive bladder medications (e.g., anti-muscarinics, beta-3-adrenergic agonists) <3 months before screening.
2. Initiation, dose escalation, or weaning of BPH medications <1 month before screening (<6 months for 5-alpha-reductase inhibitors). Participants' must also be willing to not start, stop, or change their BPH medications for the subsequent 7 months (the entire study period).
3. Initiation, dose escalation, or weaning of other pharmacologic agents or dietary supplements that might affect LUTS (e.g., saw palmetto, testosterone, diuretics, glucose-lowering agents) <1 month before screening. Participants' must also be willing to not start, stop, or change these medications for the subsequent 7 months (the entire study period) unless deemed necessary by their clinician.
4. History of BPH procedure or surgery.
5. History of overactive bladder procedure (e.g., intravesical Botox, sacral neuromodulation, posterior tibial nerve stimulation).
6. History of prostate cancer (treated with surgery or radiation), bladder cancer, other lower urinary tract cancer, pelvic radiation, or active non-urologic cancer treatments.
7. History of urethral strictures.
8. History of neurogenic bladder or neurologic conditions causing lower urinary tract dysfunction (e.g., Parkinson's disease, multiple sclerosis, other progressive neurological disease).
9. History of recurrent bladder or prostate infections (3 or more infections in the previous 12 months before screening).
10. History of severe or end-stage chronic kidney disease disease, kidney transplant, heart transplant, congenital heart disease, severe heart failure (defined as current New York Heart Association (NYHA) Class III or IV), valvular heart disease, diabetic coma, or the presence of a pacemaker or implantable cardiac defibrillator without clinician clearance.
11. Heart attack or myocardial infarction, heart surgery, cardiac catheterization, stroke, transient ischemic attack, brain hemorrhage, bleeding brain aneurysm, blood clot in leg or lungs, symptomatic hypoglycemia or hyperglycemia, hip fracture, or non-elective hospitalization <6 months before screening. If conditions occurred 6 to <12 months before screening, can participate with clinician clearance.
12. Bladder or prostate infection <1 months before screening. If infection occurred between 1 to <3 months before screening, can participate with clinician clearance.
13. Major surgery <3 months before screening or scheduled in the subsequent 7 months.
14. Terminal illness diagnosis with estimated life expectancy <12 months.
15. Plan to leave the study area for >28 consecutive days during the subsequent 7 months.
16. Participation in formal behavioral LUTS interventions (e.g., pelvic floor physiotherapy) <1 month before screening.
17. Symptoms of possible coronary artery disease, heart failure, arrythmia, stroke, carotid artery stenosis, valvular heart disease, blood clot in lungs, poorly controlled diabetes, peripheral vascular disease, or bladder or prostate infection without clinician clearance.
18. Maximum urinary flow rate <=4 ml/sec OR volume voided during free flow <120ml during screening or the baseline visit.
19. Post-void residual >=450ml measured by ultrasound during screening or the baseline visit.
20. Uncontrolled hypertension (systolic blood pressure >180mmHg or diastolic blood pressure >110mmHg) or hypotension (systolic blood pressure<100mmHg) measured during baseline visit anthropometric assessments.
21. Severe abnormalities on standard clinical labs measured prior to the baseline visit, without clinician clearance, including hemoglobin A1c (>10%) and urinary albumin: creatinine ratio (>300 mg/g).
22. Other medical, psychiatric, or behavioral factors or participation in other research studies that, based on the judgment of the multiple principal investigators, may interfere with study participation, assessments, or the ability to follow either the exercise intervention or the health education control.
23. Use of a permanent or temporary urinary catheter.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: proportion randomized | 18-24 months
  Proportion of participants randomized of those screened (completed screening call)
Acceptability: proportion satisfied with exercise intervention | 3 months
  Proportion of participants who report being satisfied or very satisfied with the exercise intervention at 12 weeks, assessed via digital survey prior to the week 12 visit
Fidelity: proportion completing at least 70% of exercise sessions | 3 months
  Proportion of intervention arm non-drop-outs completing at least 70% of exercise sessions over 12 weeks
Safety: number of adverse events | 3 months
  Number of adverse events, serious adverse events, and unexpected problems (as defined in the Data and Safety Monitoring Plan) by study. Adverse event severity will be defined by the Common Terminology Criteria for Adverse Events (CTCAE) and whether "attributable" to the exercise intervention.
Change in International Prostate Symptom Score | 3 months
  Change in International Prostate Symptom Score (IPSS) from weeks 0 to 12, collected via digital surveys prior to week 0 (baseline) and 12-week visits. Range: 0 (minimum - better) to 35 (maximum - worse)
Change in maximum urinary flow rate | 3 months
  Change in maximum urinary flow rate (Q max) from weeks 0 to 12, measured by trained clinical urology staff using a uroflowmeter in mL per second

SECONDARY OUTCOMES:
Acceptability: proportion who would recommend exercise intervention | 3 months
  Proportion of intervention arm participants who would recommend the exercise intervention to others at 12 weeks, assessed via digital survey prior to the week 12 visit
Fidelity: number of exercise sessions completed for aerobic, resistance, and balance/flexibility exercise | 3 months
  Number of exercise sessions completed over 12 weeks, recorded by the exercise coach based on participant exercise session records. The coach will also report the number of aerobic and resistance exercise sessions completed as prescribed or with greater duration or intensity (e.g., higher heart rate for aerobic sessions or greater sets, reps, and/or weight for resistance sessions) over 12 weeks, based on coaching calls.

CONTACTS AND LOCATIONS:
Overall Officials: Scott R. Bauer, MD, ScM, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - UCSF Health - Mission Bay Campus, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
As required by NIH rules, data collected as part of the proposed research will be made available to outside investigators, but within the limitations of preserving the anonymity and privacy of individuals. To maintain compliance with HIPAA regulations, our preferred method will be to execute a data sharing agreement with the requestor for a limited use dataset as defined by the US Department of Health and Human Services (DHHS). Although the investigators will require w data, the investigators propose a mechanism for sharing anonymized study data with investigators who do not choose to collaborate with the study.
Supporting Information: Analytic Code
Time Frame: After study completion
Access Criteria: Investigators will have to execute a data use agreement before documents with data from the study are sent.